CLINICAL TRIAL: NCT02614027
Title: Prevalence of Lipodystrophy Syndrome and Secondary Metabolic Syndrome in HIV-infected Patients
Brief Title: Prevalence of Lipodystrophy Syndrome and Its Role as Cause of Metabolic Disturbances
Acronym: METALIP
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Sponsor
Other Study IDs: 460/15; EC 460/15 (Other: Ethics Committee)
Record Dates: First submitted 2015-11-21; First posted 2015-11-25 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Lipodystrophy; Metabolic Syndrome
MeSH Terms: conditions — Lipodystrophy; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Evaluation of metabolic syndrome — Evaluation and analytical determinations of the different components of the syndrome
Other: Evaluation of changes in fat by DXA while on current therapy — Comparison of changes in fat (visceral and subcutaneous) by dual X-ray absorptiometry since therapy initiation

SUMMARY:
To evaluate the prevalence of lipodystrophy syndrome in patients receiving currently available antiretroviral drugs, and the prevalence of associated metabolic syndrome in HIV-infected patients with a previous diagnosis of lipodystrophy syndrome, according to the severity of fat accumulation and antiretroviral drug use.

DETAILED DESCRIPTION:
Cross-sectional evaluation of two groups of patients:

* patients receiving currently available drugs, in order to determine the changes in fat accumulation by successive dual X-ray absorptiometry (DXA) determinations
* patients with previous lipodystrophy syndrome, as evaluated by questionnaire (HOPS) and total body dual X-ray absorptiometry (DXA), in order to determine the prevalence of hypertension, low high density lipoprotein (HDL)-cholesterol, glucose disturbance (insulin resistance or diabetes), fat accumulation (waist circumference) and hypertriglyceridemia.

The prevalence of Metabolic syndrome will be evaluated according to the different definitions (IDF, NCEP-ATP III, WHO).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Older than 18 years
* Receiving first or second antiretroviral regimen or
* Previous evaluation and classification of lipodystrophy syndrome

Exclusion Criteria:

* Pregnancy
* Diagnosis of hypothyroidism, Cushing's syndrome or prolonged intake of corticosteroids or hormones before inclusion
* Patients who had received antiretroviral drugs known to produce fat disturbances (for lipodystrophy prevalence objective)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients on antiretroviral therapy with current drugs (excluding drugs previously associated with fat disturbance), and HIV-infected patients with previous evaluation of lipodystrophy syndrome in different severity, as determined by DXA and questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome as defined by the NCEP-ATP III (National Cholesterol Education Programme-Adult Treatment Panel III) | 3 months
  Prevalence of the different components of this syndrome: Abdominal obesity: waist circumference ≥102 cm in men and ≥88 cm in women, hypertriglyceridemia: ≥150 mg/dl (1.695 mmol/l), low HDL-C: <40 mg/dl in men and <50 mg/dl in women, high blood pressure (BP): >130/85 mmHg, and high fasting glucose: >110 mg/dl.
Prevalence of lipodystrophy syndrome as defined by changes in fat by DXA | 6 meses
  Comparison of changes in visceral and subcutaneous fat during current antiretroviral therapy for patients receiving current antiretroviral regimens and who never received thymidine analogues, didanosine, lopinavir, indinavir, or nelfinavir.

SECONDARY OUTCOMES:
Value of dual X-ray absorptiometry (DXA) in predicting the development of lipodystrophy and metabolic syndrome | 3 months
  Correlations of visceral fat by DXA with fat accumulation, hypertension, diabetes or hypertriglyeceridemia

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, MD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided